CLINICAL TRIAL: NCT03240094
Title: PhysioDom Home Dietary Intake Monitoring: Telemonitoring of Nutritional Parameters and Other Outcomes in Community Dwelling Elderly People: a Process and Effect Study.
Brief Title: Feasibility and Effectiveness of Nutritional Telemonitoring in Community-dwelling Elderly.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: European Union (Other); Consorci Sanitari de Terrassa (Other); Viveris Technologies SA (Unknown); STMicroelectronics Grenoble 2 SAS (Unknown); Sirlan Technologies SAS (Unknown); Habitat Health Environment (Other); Universite Paris 13 (Unknown); Meditecnologia SA (Unknown); Cybermoor Ltd (Other); Telecom Sante (Unknown); Zorggroep Noordwest-Veluwe (Other); Opella (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL53619.081.15
Record Dates: First submitted 2017-07-24; First posted 2017-08-04 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-07

CONDITIONS: Undernutrition; Aging
Keywords: Ehealth; Older adults; Undernutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional telemonitoring (Experimental): Participants in the intervention group receive a telemonitoring intervention, including self-measurements of body weight, nutritional status, appetite, diet quality, and physical activity. Additionally, participants receive guidance on nutrition and physical activity by means of customized and general television messages and/or if necessary personal guidance by a nurse.
  Interventions: Other: Nutritional telemonitoring
- Usual care (No Intervention): Participants in the control group receive usual care.

INTERVENTIONS:
Other: Nutritional telemonitoring — Participants receive a weighing scale, pedometer and television channel in order to perform self measurements and receive guidance on nutrition and physical activity. Nurses use a website in order to receive telemonitoring measurements and decide about proper follow-up. In case of risk of undernutrition, nurses provide personal advice to optimize nutritional status of the participant.
  Arms: Nutritional telemonitoring

SUMMARY:
An optimal nutritional status is essential for healthy ageing. Telemonitoring might contribute to maintaining or improving nutritional status in elderly people.The objectives of this effect study are to test the feasibility and effectiveness of telemonitoring of nutritional parameters in community-dwelling older adults.

ELIGIBILITY:
Inclusion Criteria:

Having a care referral for at least one of the following types of care:

* Domestic care
* Personal care
* Nursing care
* Individual or group support
* Living in a sheltered home or service flat

Exclusion Criteria:

* Severe cognitive impairment (Mini Mental State Examination (MMSE) < 20)
* Receiving terminal care
* Not having a television at home
* Clients with a visual impairment (not able to watch the television screen)
* Clients with a physical impairment in such a way, that they are not able to use the telemonitoring system
* Clients with nursing home care

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 213 (Actual)
Dates: Start 2016-02-26 (Actual); Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

PRIMARY OUTCOMES:
Nutritional status (MNA) | 6 months
  Measured by Mini Nutritional Assessment

SECONDARY OUTCOMES:
Behavioural determinant: Knowledge | 6 months
  Measured with 11 knowledge statements to be answered by true/false/don't know
Behavioural determinant: Goalsetting | 6 months
  Measured by three items to be answered on a 5 point likert scale on a 5-point likert scale.
Behavioural determinant: Intention to eat healthy | 6 months
  Measured by three items to be answered on a 5 point likert scale on a 5-point likert scale.
Behavioural determinant: Intention to improve physical activity | 6 months
  Measured by three items to be answered on a 5 point likert scale on a 5-point likert scale.
Behavioural determinant: Self efficacy | 6 months
  Measured by two items to be answered on a 5 point likert scale on a 5-point likert scale.
Behavioural determinant: Perceived behavioural control | 6 months
  Measured by five items to be answered on a 5 point likert scale on a 5-point likert scale.
Behavioural determinants: Attitude | 6 months
  Measured by 14 items to be answered on a 5 point likert scale
Diet quality (DHD-index) | 6 months
  Measured by Dutch Healthy Diet index (DHD-index)
Appetite (SNAQ) | 6 months
  Measured by Simplified Nutritional Appetite Questionnaire
Body weight (kg) | 6 months
  Measured by weighing scale of the brand A&D, type UC-411PBT-C
Physical functioning (SPPB) | 6 months
  Measured by Short Physical Performance Battery (SPPB)
Functional status (KATZ-15) | 6 months
  Measured by KATZ-15
Quality of life (SF-36) | 6 months
  Measured by Short-Form 36

CONTACTS AND LOCATIONS:
Overall Officials: Lisette de Groot, Professor, Study Chair — Wageningen University & Research; Marije van Doorn, MSc, Principal Investigator — Wageningen University & Research; Jeanne de Vries, PhD, Principal Investigator — Wageningen University & Research; Annemien Haveman, PhD, Principal Investigator — Wageningen University & Research
Locations (1):
- Wageningen University & Research, Wageningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Doorn-van Atten MN, Haveman-Nies A, Pilichowski P, Roca R, de Vries JHM, de Groot CPGM. Telemonitoring to improve nutritional status in community-dwelling elderly: design and methods for process and effect evaluation of a non-randomized controlled trial. BMC Geriatr. 2018 Nov 16;18(1):284. doi: 10.1186/s12877-018-0973-2. PMID 30445922
- [Derived] van Doorn-van Atten MN, Haveman-Nies A, van Bakel MM, Ferry M, Franco M, de Groot LCPGM, de Vries JHM. Effects of a multi-component nutritional telemonitoring intervention on nutritional status, diet quality, physical functioning and quality of life of community-dwelling older adults. Br J Nutr. 2018 May;119(10):1185-1194. doi: 10.1017/S0007114518000843. PMID 29759110